CLINICAL TRIAL: NCT03702413
Title: Randomized Controlled Trial of Endovascular Therapy for Acute Large Vessel Occlusion With Large Ischemic Core (RESCUE Japan LIMIT)
Brief Title: Randomized Controlled Trial of Endovascular Therapy for Acute Large Vessel Occlusion With Large Ischemic Core
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hyogo Medical University (Other)
Responsible Party: Principal Investigator, Shinichi Yoshimura, Department of Neurosurgery, Hyogo Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R000038184
Record Dates: First submitted 2018-10-04; First posted 2018-10-11 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Mechanical Thrombectomy; Large Ischemic Core
Keywords: Acute cerebral infarction due to large vessel occlusion; Mechanical thrombectomy; Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Best medical treatment (No Intervention): Best medical treatment
- Endovascular treatment (Experimental): Best medical treatment plus endovascular treatment
  Interventions: Procedure: Endovascular treatment

INTERVENTIONS:
Procedure: Endovascular treatment — Acute thrombectomy
  Arms: Endovascular treatment

SUMMARY:
RESCUE-Japan LIMIT(Recovery by Endovascular Salvage for Cerebral Ultra-acute Embolism Japan Large IscheMIc core Trial) is a prospective, open label, blinded endpoint (PROBE), Japanese, two-arm, randomized, controlled, post-market study to compare the effectiveness of endovascular treatment as compared to best medical treatment alone in the acute ischemic stroke patients with an low ASPECTS (CT-ASPECTS 3-5 or DWI-ASPECTS 3-5).

The purpose of this study is to investigate the efficacy of endovascular treatment for acute large vessel occlusion with large ischemic core (CT-ASPECT score 3-5 or DWI-ASPECT score 3-5).

DETAILED DESCRIPTION:
In the American Heart Association guideline 2018, endovascular therapy (EVT) has been strongly recommended as class of recommendation (COR) I for for the patients with acute cerebral large vessel occlusion (LVO), the Alberta Stroke Program Early CT Score (ASPECTS) 6 or more. The efficacy of EVT for the patients with low ASPECTS remains unclear.

This study is a prospective, open label, blinded endpoint (PROBE), Japanese, two-arm, randomized, controlled, post-market study to compare the effectiveness of endovascular treatment as compared to best medical treatment alone for acute large vessel occlusion patients with large ischemic core (ASPECTS 3-5 or DWI-ASPECTS 3-5).

Up to 200 subjects will be enrolled in the study and randomized for the Intention to treat analysis set. The randomization will be stratified by treatment institutes, patient's age (less than 75 years old or not), time from symptom onset (0-2 hours or more than 2 hours), and stroke severity (NIHSS 21 or more/less than 21), and administration of rt-PA.

Subjects who meet the inclusion criteria will be randomized in a 1:1 ratio to one of the following two treatment arms: Arm 1: best medical treatment Arm 2: best medical treatment plus endovascular treatment

Primary outcome of this study is to investigate efficacy of endivascular treatment in acute stroke patients with large ischemic core (ASPECTS 3-5 or DWI-ASPECTs 3-5) as compared to best medical treatment alone.

Approximately 40 sites in Japan Patients presenting with acute ischemic stroke (AIS) based on focal occlusion in the M1 segment of the middle cerebral artery (MCA), and/or the intracranial segment of the distal internal carotid artery (ICA), determined by Magnetic Resonance Angiography (MRA) or Computed Tomographic Angiography (CTA), and who meet all eligibility criteria will be considered for study enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Acute cerebral infarction
2. Age ≥ 18
3. NIHSS ≥ 6
4. Prestroke Modified Rankin Score 0-1
5. ICA or M1 Occlusion on CT angiography or MR angiography
6. ASPECTS 3-5 or DWI-ASPECTS 3-5
7. Randamization can be finished within 6 hours from last known well time, or 6 to 24 hours from last well known well time without positive lesion on MRI-FLAIR image.
8. Endovascular treatment can be initiatedwithin 60 minutes from randomization
9. Patient or Legally Authorized Representative has signed the Informed Consent form

Exclusion Criteria:

1. Significant mass effect with midline shift
2. Known allergy to contrast agents
3. Evidence of acute intracranial hemorrhage
4. Female who is pregnant or suspicision of pregnant
5. Clinical evidence of chronic occlusion
6. High risk of hemorrhage (platelet < 40,000 /µL, APTT > 50 second or PT-INR > 3.0)
7. Participating in any other therapeutic investigational trial
8. Subjects who, in the judgment of the investigator, are likely to be non-compliant or uncooperative during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale ≤3 at 90 days | 90 days
  The primary endpoint of the trial is the modified Rankin Scale (mRS) ≤3 at 90 days post-stroke.The scale runs from 0-6 with 0 being perfect health without symptoms to 6 being death.
  0: No symptoms.
  1. No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. Slight disability. Able to look after own a符airs without assistance, but unable to carry out all previous activities.
  3. Moderate disability. Requires some help, but able to walk unassisted.
  4. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. Severe disability. Requires constant nursing care and a悦ention, bedridden, incontinent.
  6. Dead.

SECONDARY OUTCOMES:
modified Rankin Scale≤2 at 90 days | 90 days
  Functional independence as difined by modified Rankin ScalemRS≤2 at 90 days
modified Rankin Scale≤1 at 90 days | 90 days
  Excellent outcome as difined by modified Rankin Scale≤1 at 90 days
Distribution of patients across the ordinal modified Rankin scale | 90 days
  The difference in linear trends in ordinal mRS outcomes between treatment groups (mRS shift analysis)
NIHSS improvement 8 points or more at 48 hours | 48 hours
  Early improvement of neulogical findings
Symptomatic intracranial hemorrhage within 48 hours | 48 hours
  Defined as NIHSS worsening of 4 or more points associated with ICH within 48 hours of randomization
Intracranial hemorrhage within 48 hours | 48 hours
  The incidence of hemorrhage
Death | 90 days
  Death due to any cause at 90 days
Recurrence of cerebral infarction within 90 days | 90 days
  Recurrence of cerebral infarction
Propotion of subjects who required decompressive craniectomy within 7 days | 7 days
  Propotion of subjects who had space-occupying infarction (malignant brain edema) and requred decompressive craniectomy within 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Shinichi Yoshimura, phD, Study Chair — Hyogo Medical University
Locations (1):
- Hyogo collage of Medicine, Nishinomiya, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanaka K, Yoshimoto T, Koge J, Yamagami H, Imamura H, Sakai N, Uchida K, Beppu M, Matsumaru Y, Matsumoto Y, Kimura K, Ishikura R, Inoue M, Sakakibara F, Morimoto T, Yoshimura S, Toyoda K; RESCUE-Japan LIMIT Investigators. Detrimental Effect of Acute Hyperglycemia on the Outcomes of Large Ischemic Region Stroke. J Am Heart Assoc. 2024 Dec 3;13(23):e034556. doi: 10.1161/JAHA.124.034556. Epub 2024 Nov 22. PMID 39575760
- [Derived] Inoue M, Yoshimoto T, Yamagami H, Toyoda K, Sakai N, Matsumaru Y, Matsumoto Y, Kimura K, Ishikura R, Uchida K, Beppu M, Sakakibara F, Morimoto T, Yoshimura S; RESCUE-Japan LIMIT Investigators. Expanding the Treatable Imaging Profile in Patients With Large Ischemic Stroke: Subanalysis From a Randomized Clinical Trial. Stroke. 2024 Jul;55(7):1730-1738. doi: 10.1161/STROKEAHA.124.046828. Epub 2024 May 28. PMID 38804134
- [Derived] Shindo S, Uchida K, Yoshimura S, Sakai N, Yamagami H, Toyoda K, Matsumaru Y, Matsumoto Y, Kimura K, Ishikura R, Inoue M, Sakakibara F, Nakajima M, Ueda M, Morimoto T. Intravenous alteplase before endovascular therapy for acute large vessel occlusion with large ischemic core: subanalysis of a randomized clinical trial. J Neurointerv Surg. 2024 Oct 14;16(11):1094-1100. doi: 10.1136/jnis-2023-020846. PMID 37890987
- [Derived] Ospel JM, Kunz WG, McDonough RV, Goyal M, Uchida K, Sakai N, Yamagami H, Yoshimura S; RESCUE-Japan LIMIT Investigators. Cost-effectiveness of Endovascular Treatment for Acute Stroke with Large Infarct: A United States Perspective. Radiology. 2023 Oct;309(1):e223320. doi: 10.1148/radiol.223320. PMID 37787675
- [Derived] Namitome S, Uchida K, Shindo S, Yoshimura S, Sakai N, Yamagami H, Toyoda K, Matsumaru Y, Matsumoto Y, Kimura K, Ishikura R, Inoue M, Beppu M, Sakakibara F, Shirakawa M, Ueda M, Morimoto T; RESCUE-Japan LIMIT Investigators. Number of Passes of Endovascular Therapy for Stroke With a Large Ischemic Core: Secondary Analysis of RESCUE-Japan LIMIT. Stroke. 2023 Aug;54(8):1985-1992. doi: 10.1161/STROKEAHA.123.042552. Epub 2023 Jul 7. PMID 37417239
- [Derived] Uchida K, Shindo S, Yoshimura S, Toyoda K, Sakai N, Yamagami H, Matsumaru Y, Matsumoto Y, Kimura K, Ishikura R, Yoshida A, Inoue M, Beppu M, Sakakibara F, Shirakawa M, Morimoto T; RESCUE-Japan LIMIT Investigators. Association Between Alberta Stroke Program Early Computed Tomography Score and Efficacy and Safety Outcomes With Endovascular Therapy in Patients With Stroke From Large-Vessel Occlusion: A Secondary Analysis of the Recovery by Endovascular Salvage for Cerebral Ultra-acute Embolism-Japan Large Ischemic Core Trial (RESCUE-Japan LIMIT). JAMA Neurol. 2022 Dec 1;79(12):1260-1266. doi: 10.1001/jamaneurol.2022.3285. PMID 36215044
- [Derived] Yoshimura S, Sakai N, Yamagami H, Uchida K, Beppu M, Toyoda K, Matsumaru Y, Matsumoto Y, Kimura K, Takeuchi M, Yazawa Y, Kimura N, Shigeta K, Imamura H, Suzuki I, Enomoto Y, Tokunaga S, Morita K, Sakakibara F, Kinjo N, Saito T, Ishikura R, Inoue M, Morimoto T. Endovascular Therapy for Acute Stroke with a Large Ischemic Region. N Engl J Med. 2022 Apr 7;386(14):1303-1313. doi: 10.1056/NEJMoa2118191. Epub 2022 Feb 9. PMID 35138767